CLINICAL TRIAL: NCT06534424
Title: The caRe Study: Clinical Application of Refined Risk Estimates
Brief Title: Clinical Impact of Enhanced Risk Assessments in Women With a BRCA1/2 Mutation, CARE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Amanda Toland, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-17057; NCI-2022-07731 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: BRCA1/2-Associated Hereditary Breast and Ovarian Cancer Syndrome
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Counseling; Genotype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (enhanced risk assessment) (Experimental): Patients undergo collection of blood or mouthwash samples. Patients undergo genotyping with enhanced risk assessment on study. 4 to 8 weeks later, patients receive a follow-up phone call for return of enhanced risk assessment results and tailored counseling.
  Interventions: Procedure: Biospecimen Collection; Other: Counseling; Procedure: Discussion; Procedure: Genotyping; Procedure: Molecular Risk Assessment; Other: Questionnaire Administration
- Arm II (standard) (Active Comparator): Patients undergo collection of blood or mouthwash samples. 4-8 weeks later, patients receive a standard follow-up phone call.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Discussion; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard)
Procedure: Biospecimen Collection — Undergo collection of blood or mouthwash sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Counseling — Receive tailored counseling
  Other Names: Counseling Intervention
  Arms: Arm I (enhanced risk assessment)
Procedure: Discussion — Participate in phone discussion
  Other Names: Discuss
Procedure: Genotyping — Undergo genotyping
  Other Names: GENOTYPE; Genotype Analysis; Genotype Assay
  Arms: Arm I (enhanced risk assessment)
Procedure: Molecular Risk Assessment — Undergo enhanced risk assessment
  Arms: Arm I (enhanced risk assessment)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the impact of enhanced risk assessments on knowledge, perceptions, and decisional conflict about cancer prevention in women with a BRCA1 or BRCA2 mutation. BRCA1/2 mutation carriers have a much higher risk of developing breast and ovarian cancer. Due to the high risk of cancer, mutation carriers are provided guidelines on more intensive screening and preventative surgeries such as bilateral mastectomy and bilateral salpingo-oophorectomy. Doctors want to learn if a more personalized risk assessment impacts the patients' risk perceptions and comfort with decision-making around cancer prevention behaviors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To deploy tools for delivering enhanced genetic risk predictions based on BRCA1/2 genetic risk modifiers in a clinical setting and assess the impact of risk stratification on genetic knowledge, risk perceptions and decisional conflict regarding cancer prevention decision-making.

II. To perform long-term follow-up of individuals in the randomized controlled trial (RCT) to determine if there are differences in satisfaction, decision-making and outcomes in individuals who received standard versus enhanced genetic risk predictions over time.

OUTLINE: Patients undergo collection of blood or mouthwash samples. Patients are then randomized to 1 of 2 arms.

ARM I: Patients undergo genotyping with enhanced risk assessment on study. 4 to 8 weeks later, patients receive a follow-up phone call for return of enhanced risk assessment results and tailored counseling.

ARM II: 4-8 weeks later, patients receive a standard follow-up phone call.

After completion of study intervention, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have had genetic counseling and testing for mutations in BRCA1 and/or BRCA2 through a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* Were found to have a known pathogenic mutation upon testing
* Are within 3 weeks of results disclosure
* Have available medical records for ascertainment of clinical information
* Are able to provide a source of deoxyribonucleic acid (DNA) (blood or mouthwash) for study
* Have access to a telephone and a computer or other internet-ready device
* Have not yet had a bilateral prophylactic mastectomy or bilateral Salpingo oophorectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Decisional conflict Regarding Cancer Risk Management | Up to 3 months
  Decisional conflict regarding cancer risk management will be measured via a questionnaire. Comparison of this measure between the enhanced and standard arms adjusting for stratified randomization will be made using linear regression. The alpha level for the outcome will be 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Toland, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu